CLINICAL TRIAL: NCT00135551
Title: The Combination Therapy of Hypertension to Prevent Cardiovascular Events Trial
Brief Title: Benidipine-based Comparison of Angiotensin Receptors, β-blockers, or Thiazide Diuretics in Hypertensive Patients
Acronym: COPE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Seiji Umemoto, M.D., Ph.D. (Other)
Collaborators: The Japanese Society of Hypertension (Other); Yamaguchi University Hospital (Other); Kyowa Hakko Kogyo Co., Ltd. (Industry)
Responsible Party: Sponsor-Investigator, Seiji Umemoto, M.D., Ph.D., Associate Professor, COPE Trial Group
Organization: COPE Trial Group (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: copeadministrator
Record Dates: First submitted 2005-08-24; First posted 2005-08-26 (Estimated); Last update posted 2012-02-22 (Estimated); Status verified 2012-02

CONDITIONS: Cardiovascular Disease
Keywords: Hypertension; Multicenter clinical trial; PROBE; Combination therapy; Benidipine; Essential Hypertension
MeSH Terms: conditions — Cardiovascular Diseases; Hypertension; Essential Hypertension | interventions — Angiotensin Receptor Antagonists; benidipine; Sodium Chloride Symporter Inhibitors

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- angiotensin receptor blockers (Active Comparator): benidipine+angiotensin receptor blockers, titlation scheme
  Interventions: Drug: Angiotensin receptor blockers
- β-blockers (Active Comparator): benidipie+β-blockers, titlation scheme
  Interventions: Drug: β-blockers
- thiazide diuretics (Active Comparator): benidipine+thiazide diuretics, titlation scheme
  Interventions: Drug: thiazide diuretics

INTERVENTIONS:
Drug: Angiotensin receptor blockers — benidipine+angiotensin receptor blocker, titlation scheme
  Other Names: benidipine, angiotensin receptor blockers
  Arms: angiotensin receptor blockers
Drug: β-blockers — benidipine+β-blockers, titlation scheme
  Other Names: benidipine, β-blockers
  Arms: β-blockers
Drug: thiazide diuretics — benidipie+thiazide diuretics, titlation scheme
  Other Names: benidipie, thiazide diuretics
  Arms: thiazide diuretics

SUMMARY:
A number of major clinical trials have demonstrated the clinical benefits of lowering blood pressure and have indicated that a majority of patients with hypertension will require more than one drug to achieve optimal blood pressure control.

There is little data showing which antihypertensive combination best protects patients from cardiovascular events and which best achieves the target blood pressure with the fewest adverse events.

The COPE trial is planned to investigate, in patients with hypertension, which combination of the antihypertensive drugs, angiotensin receptor blockers, β-blockers or thiazide diuretics in addition to a long-acting calcium antagonist, benidipine hydrochloride, is superior to achieve the targeted blood pressure and prevent cardiovascular events with the fewest adverse drug effects.

ELIGIBILITY:
Inclusion Criteria:

* Outpatients who are required a combination therapy with sitting systolic blood pressure ≥ 140 mmHg or diastolic blood pressure ≥ 90 mmHg.
* Outpatients aged over 40 years and less than 85 years (inclusive), regardless of sex.
* Previously untreated patients or patients who are on other therapy, which can be converted to 4mg of benidipine.
* Patients who can be treated with benidipine, angiotensin receptor blockers, β-blockers, and thiazide diuretics.

Exclusion Criteria:

* Seated systolic blood pressure ≥ 200 mmHg or seated diastolic blood pressure ≥ 120 mmHg.
* Secondary hypertension.
* Type I diabetes mellitus or type 2 diabetes on insulin treatment.
* History of cerebrovascular disorder, myocardial infarction, angina pectoris, coronary angioplasty or coronary artery bypass graft surgery within 6 months prior to enrolment in the study.
* Heart failure (New York Heart Association [NYHA] functional classification II, III or IV).
* Chronic atrial fibrillation or atrial flutter.
* Congenital heart disease or a history of rheumatic heart disease.
* Severe peripheral arterial disease (Fontaine Class II, III or IV).
* Serious liver dysfunction (AST or ALT ≥100 IU / l).
* Serious renal dysfunction (serum creatinine ≥ 2mg/dl).
* History of malignancy 5 years prior to study entry.
* Pregnancy.
* Compliance rate < 70% assessed by a patient interview.
* Known hypersensitivity or contraindication to benidipine, angiotensin receptor blockers, β-blockers, and thiazide diuretics.
* Other serious illness or significant abnormalities that the investigator judges inappropriate for the study

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3501 (Actual)
Dates: Start 2003-05; Primary Completion 2010-05 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
A composite of fatal and non-fatal cardiovascular events. | first event
Achievement of target blood pressure (< 140 mmHg/90 mmHg). | time course

SECONDARY OUTCOMES:
All-cause mortality. | first event
Death from cardiovascular events. | first event
Fatal and non-fatal cardiovascular events. | first event
Hospitalization due to heart failure. | first event
New onset of diabetes mellitus. | first event
Safety (adverse events and adverse drug reaction). | total number

CONTACTS AND LOCATIONS:
Overall Officials: Toshio Ogihara, MD, PhD, Principal Investigator — Department of Geriatric Medicine, Osaka University Graduate School of Medicine; Takao Saruta, MD, PhD, Study Chair — Department of Internal Medicine, Keio University School of Medicine
Locations (1):
- Department of Medicine and Clinical Science, Yamaguchi University Graduate School of Medicine, Ube, Yamaguchi, Japan

REFERENCES:
- [Background] Ogihara T, Matsuzaki M, Matsuoka H, Shimamoto K, Shimada K, Rakugi H, Umemoto S, Kamiya A, Suzuki N, Kumagai H, Ohashi Y, Takishita S, Abe K, Saruta T; COPE Trial Group. The combination therapy of hypertension to prevent cardiovascular events (COPE) trial: rationale and design. Hypertens Res. 2005 Apr;28(4):331-8. doi: 10.1291/hypres.28.331. PMID 16138563
- [Result] Matsuzaki M, Ogihara T, Umemoto S, Rakugi H, Matsuoka H, Shimada K, Abe K, Suzuki N, Eto T, Higaki J, Ito S, Kamiya A, Kikuchi K, Suzuki H, Tei C, Ohashi Y, Saruta T; Combination Therapy of Hypertension to Prevent Cardiovascular Events Trial Group. Prevention of cardiovascular events with calcium channel blocker-based combination therapies in patients with hypertension: a randomized controlled trial. J Hypertens. 2011 Aug;29(8):1649-59. doi: 10.1097/HJH.0b013e328348345d. PMID 21610513
- [Result] Ogihara T, Matsuzaki M, Umemoto S, Rakugi H, Matsuoka H, Shimada K, Higaki J, Ito S, Kamiya A, Suzuki H, Ohashi Y, Shimamoto K, Saruta T; Combination Therapy of Hypertension to Prevent Cardiovascular Events Trial Group. Combination therapy for hypertension in the elderly: a sub-analysis of the Combination Therapy of Hypertension to Prevent Cardiovascular Events (COPE) Trial. Hypertens Res. 2012 Apr;35(4):441-8. doi: 10.1038/hr.2011.216. Epub 2012 Jan 26. PMID 22278623
- [Derived] Umemoto S, Ogihara T, Matsuzaki M, Rakugi H, Shimada K, Hayashi K, Makino H, Ohashi Y, Saruta T. Effects of an Antihypertensive Combination in Japanese Hypertensive Outpatients Based on the Long-acting Calcium Channel Blocker Benidipine on Vascular and Renal Events: A Sub-analysis of the COPE Trial. Curr Hypertens Rev. 2020;16(3):238-245. doi: 10.2174/1573402116666200129130151. PMID 31995012
- [Derived] Umemoto S, Ogihara T, Matsuzaki M, Rakugi H, Ohashi Y, Saruta T; Combination Therapy of Hypertension to Prevent Cardiovascular Events COPE Trial Group. Effects of calcium channel blocker-based combinations on intra-individual blood pressure variability: post hoc analysis of the COPE trial. Hypertens Res. 2016 Jan;39(1):46-53. doi: 10.1038/hr.2015.104. Epub 2015 Oct 22. PMID 26490089
- [Derived] Umemoto S, Ogihara T, Rakugi H, Matsumoto M, Kitagawa K, Shimada K, Higaki J, Ito S, Suzuki H, Ohashi Y, Saruta T, Matsuzaki M; Combination Therapy of Hypertension to Prevent Cardiovascular. Effects of a benidipine-based combination therapy on the risk of stroke according to stroke subtype: the COPE trial. Hypertens Res. 2013 Dec;36(12):1088-95. doi: 10.1038/hr.2013.100. Epub 2013 Aug 29. PMID 23985703
- See also: Japanese Society of Hypertension — http://www.jpnsh.org/index_e.html
- See also: Department of Geriatric Medicine, Osaka University Graduate School of Medicine — http://www.med.osaka-u.ac.jp/pub/geriat/www/